CLINICAL TRIAL: NCT01863888
Title: Exploratory Open Label Study to Investigate the Effect of Teriflunomide on Immune Cell Subsets in the Blood of Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Effect of Teriflunomide on Immune Cell Subsets in the Blood of Patients With Multiple Sclerosis
Acronym: TERI-DYNAMIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS13539; U1111-1139-8802 (Other: UTN)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Cholestyramine Resin; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- teriflunomide (HMR1726) (Experimental): Participants administered 14mg Teriflunomide once daily, oral. For participants who permanently discontinue Teriflunomide, an accelerated elimination procedure with either cholestyramine or charcoal will be administered.
  Interventions: Drug: teriflunomide HMR1726; Drug: cholestyramine; Drug: charcoal
- Reference population (No Intervention): Untreated healthy subjects

INTERVENTIONS:
Drug: teriflunomide HMR1726 — Pharmaceutical form:tablet Route of administration: oral
  Arms: teriflunomide (HMR1726)
Drug: cholestyramine — Pharmaceutical form:powder Route of administration: oral
  Arms: teriflunomide (HMR1726)
Drug: charcoal — Pharmaceutical form:granule Route of administration: oral
  Arms: teriflunomide (HMR1726)

SUMMARY:
Primary Objective:

To measure the effect of Teriflunomide on lymphocytes subsets in patients with relapsing forms of multiple sclerosis as compared with baseline values and those of a reference population of untreated healthy subjects.

Secondary Objectives:

To assess if Teriflunomide treatment results in biased T cell clonal diversity. To assess the effect of Teriflunomide on the function of peripheral blood mononuclear cells (proliferation and cytokine production in situ).

To assess the circulating cytokines profile in the serum of Relapsing Multiple Sclerosis (RMS) patients during a 24-week treatment versus baseline and healthy controls.

To assess the reversibility of all parameter changes in patients who discontinue treatment after accelerated elimination procedure with cholestyramine or activated charcoal.

DETAILED DESCRIPTION:
The duration of the study for patients is 32 weeks which includes 4 weeks for screening, 24 weeks for treatment and 4 weeks for follow-up. An extension of the study is proposed until Teriflunomide is commercially available in the country where patient lives.

The duration of the study for healthy volunteers is 25 weeks which includes only one week for screening.

ELIGIBILITY:
Inclusion criteria:

Patients (male and female) with relapsing forms of multiple sclerosis meeting McDonald criteria for MS at the screening visit and having either one of the following treatment status:

* Naïve to disease modifying (DM) treatment or no DM treatment for more than 2 years
* Or currently (not more than 3 months interruption) on MS therapy with IFN β-1 or Glatiramer acetate and a period of at least 2 weeks without IFN β-1 or Glatiramer acetate before switching to teriflunomide.

Male and female patients, between 18 and 56 years of age, exclusive.

Healthy volunteers:

Male and female subjects, between 18 and 56 years of age, exclusive. Body weight between 50.0 and 95.0 kg, inclusive, if male; and between 40.0 and 85.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.

Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

Normal vital signs after 10 minutes resting in supine position:

* 95 mmHg < systolic blood pressure (SBP) <140 mmHg
* 45 mmHg < diastolic blood pressure (DBP) <90 mmHg
* 40 bpm < heart rate (HR) <100 bpm Normal standard 12-lead electrocardiogram (ECG) after 10 minutes resting in supine position; 120 ms < PR <220 ms, QRS <120 ms, QTc ≤ 430 ms if male, ≤ 450 ms if female.

Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for healthy subjects; however liver function parameter(s) should not exceed the upper laboratory norm.

Exclusion criteria:

Did not consent to HIV testing (the specifics of informed consent process for the HIV testing should be done in accordance with local guidelines).

A relapse within 30 days prior to screening. Clinically relevant cardiovascular, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the patient at risk by participating in the study.

Patients with a congenital or acquired severe immunodeficiency, a history of cancer (except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis), lymphoproliferative disease, or any patient who has received lymphoid irradiation.

Human immunodeficiency virus (HIV) positive patients. Known history of active tuberculosis not adequately treated or positive QuantiFERON TB Gold test.

Hypoproteinemia (eg, in case of severe liver disease or nephrotic syndrome) with serum albumin <3.0 g/dL.

Moderate to severe impairment of renal function, as shown by serum creatinine >133 μmol/L (or >1.5 mg/dL).

Patients with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia.

Acute or chronic infection. Liver function impairment or persisting elevations >1.5ULN (confirmed by retest) of serum glutamic pyruvic transaminase/ alanine aminotransferase (SGPT/ALT), serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST), or direct bilirubin greater than 1.5-fold the upper limit of normal.

Use of adrenocorticotrophic hormone (ACTH) or systemic corticosteroids for 2 weeks prior to screening.

Prior or concomitant use of cytokine therapy or intravenous immunoglobulins in the 3 months prior to screening.

Prior use of alemtuzumab or cladribine. Prior use (within 1 year) of fingolimod (Gylenia®). Prior use (within 2 years) of mitoxantrone, natalizumab (Tysabri®), or immunosuppressant agents (i.e. azathioprine, cyclophosphamide, cyclosporin, methotrexate or mycophenolate).

Prior treatment with teriflunomide, and prior or concomitant use of leflunomide (ARAVA®) or hypersensitivity to any of the other ingredients or excipients of the investigational product.

Prior use of any investigational drug in the 6 months preceding screening. Pregnant or breast-feeding women. Women of childbearing potential not utilizing effective contraceptive method and /or women of childbearing potential who are unwilling to or unable to be tested for pregnancy.

Known history of hypersensitivity to teriflunomide or leflunomide. Persisting elevations (confirmed by retest) of serum amylase or lipase greater than 2-fold the upper limit of normal.

Known history of chronic pancreatic disease or pancreatitis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Lymphocyte subset parameters as measured by flow cytometry | At 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Change from baseline in biased T cell clonal repertoire based T cell receptor (TCR) spectratyping | At 12 weeks and 24 weeks
Change from baseline in serum cytokine as measured by multicytokine array tool | At 12 weeks and 24 weeks
Change from baseline in Mitogen/TCR-specific T cell proliferation as measured by flow cytometry | At 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Belgium (3):
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056002, Overpelt
  - Investigational Site Number 056003, Sijsele-Damme
- Germany (6):
  - Investigational Site Number 276-003, Bad Mergentheim
  - Investigational Site Number 276-004, Hanover
  - Investigational Site Number 276-005, Marburg
  - Investigational Site Number 276-007, Mönchengladbach
  - Investigational Site Number 276-001, Münster
  - Investigational Site Number 276-002, Ulm
- Investigational Site Number 528001, Sittard-Geleen, Netherlands